CLINICAL TRIAL: NCT04840017
Title: The Influence of Rehabilitation Program on Postural Control, Balance and Basic Gait Parameters on the Formation of the Foot's Longitudinal Arch in Children With Flatfoot and Excessive Body Mass
Brief Title: The Influence of Rehabilitation Program on Postural Control, Balance and Gait in Children With Flatfoot
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gdansk UPES
Record Dates: First submitted 2021-02-03; First posted 2021-04-09 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-08

CONDITIONS: Flatfoot
Keywords: Planovalgus; Medial Longitudinal Arch; Gait; Kinematic; Emg; Walk; Locomotion; Motion Analysis; Low-arched Feet; Valgus Deformity; Balance
MeSH Terms: conditions — Flatfoot | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group I (Experimental): excessive body weight and flat feet
  Interventions: Other: rehabilitation exercise
- Study group II (Experimental): normal body weight and flat feet
  Interventions: Other: rehabilitation exercise
- Study group III (No Intervention): control, healthy children

INTERVENTIONS:
Other: rehabilitation exercise — Rehabilitation exercise of intrinsic foot muscles
  Arms: Study group I; Study group II

SUMMARY:
"Idiopathic flat foot is a common condition in children and adolescents. After loading, the heel is adjusted in valgus, the medial longitudinal arch of the foot flattens, and the forefoot is positioned at abducted. Such deformation can be classified as flexible or rigid. A lowered flat foot arch is an undesirable feature.

Additional factors such as e.g. abnormal body weight, may have impact on the shape of medial longitudinal arch. Increasing evidence suggests that excess weight is inextricably linked to flatfoot and postural stability.

In connection with consequences, disorders of the muscles responsible for stabilizing the arches of the foot are noticed.

The mobility and stability of the foot arches is controlled by the internal and external muscles of the foot, but the former are often overlooked in therapy. Short foot exercises are recommended as an improvement in foot arch parameters. The participants will take part in the research with the written consent of their parents or legal guardians. The results will be used anonymously for scientific publications."

DETAILED DESCRIPTION:
"Idiopathic flat foot is a common condition in children and adolescents. After loading, the heel is adjusted in valgus, the medial longitudinal arch of the foot flattens, and the forefoot is positioned at abducted. Such deformation can be classified as flexible or rigid. The importance of shaping the longitudinal arch of the foot is one of the most controversial issues in orthopedics. A lowered flat foot arch is an undesirable feature.

The shape of the arch is determined by age and genetic conditions. The age of six is believed to be a critical moment for the development of the medial longitudinal arch, since it is the age when the development of the medial longitudinal foot arch slows down to finally stop at the age of 12-13. Therefore, it seems important to pay attention to the development of the medial longitudinal arch before adolescence in order to reduce the risk of perpetuating anomalies.

Incorrect arching can cause changes in the ankle, and pronative positioning of the foot influences the adjacent joints of the lower limb and the spine, which results in impaired control of body posture, kinetics and gait kinematics. The pain induced by the changes in body functioning increases the risk of injury.

The foot is the most distal segment of the lower limb bio-kinematic chain and represents a relatively small support base while maintaining balance. Even very small changes in this segment may be the reason of disturbances in posture control strategy. In addition, elimination of longitudinal arch of the foot and hypermobile metatarsus can be a challenge for neuromuscular system in terms of stabilization and maintenance of an upright posture. When medial longitudinal arch of the foot lowers it causes functional and consequently structural disturbances. Subsequently the ability to absorb impacts decreases and the feeling of balance can be lost leading to reduced stability

There are two reasons for the adverse effects of flat foot during gait:

1. Flat feet have a shortened lever arm compared to those with correct arches. Shortening lever arm is caused by abducted forefoot in the transverse plane, hindfoot valgus and metatarsal disturbances in the sagittal plane;
2. The lever (foot) becomes more elastic due to disturbances in the metatarsal and lowering of longitudinal arch in the sagittal plane. Because of loss of an appropriate degree of lever stiffness, the energy produced by the muscles in the push-off phase is not properly used.

Additional factors such as e.g. abnormal body weight, may have impact on the shape of medial longitudinal arch. The belief that overweight or obese children have flatter feet is based on research findings and may seem like an intuitive observation. Increasing evidence suggests that excess weight is inextricably linked to flatfoot and postural stability. Excessive body weight leads to a greater overall load, with a disproportionate effect on the midfoot area and the medial longitudinal arch. Childhood overweight and obesity are not compensated by the musculoskeletal system. Weight gain imposes additional biomechanical restrictions. Evans and coauthors demonstrated the existence of a correlation between the formation of the foot arch and body weight. According to Shiang and coauthors, flat feet of obese children may be the result of a decrease in the medial longitudinal arch due to overload, which is the result of overweight. Another consequence of abnormal weight can be balance disorders. Deforche et al. proved that overweight boys show reduced ability to perform tasks requiring static and dynamic balance. Comparative studies conducted using the Y Balance Test show differences in the range of forward movement of the lower limb, to the detriment of children with abnormal body weight, which is confirmed by studies on the correlation between postural stability and excessive body weight. In connection with the above-mentioned consequences, disorders of the muscles responsible for stabilizing the arches of the foot are noticed. Similar observations were made by Sung and coauthors and Murley and coauthors showing neuromuscular compensation associated with overloading medial longitudinal arch.

The mobility and stability of the foot arches is controlled by the internal and external muscles of the foot, but the former are often overlooked in therapy. The possibility of isolated internal muscle tension of the foot is provided by ""short foot exercises"". Internal foot muscle training can improve foot function. Four-week training in adults with reduced foot arches, assessed by measuring the height of the navicular bone tuberosity and arch height index, improved balance. The results of the foot maneuver shortening test on children show that it is an effective method for increasing the arch and results in an improvement in the arch index. Short foot exercises are recommended as an improvement in foot arch parameters. Based on a meta-analysis carried out by Evans in 2008, it is believed that in the treatment of asymptomatic corrective flat feet and in disorders of their development in relation to the child's age, conservative treatment should be applied, including exercises to strengthen the intrinsic muscles of the feet. The participants will take part in the research with the written consent of their parents or legal guardians. The results will be used anonymously for scientific publications.

Hypothests: A six-week rehabilitation program for children with flat feet and excessive body weight will significantly affect the formation of the medial longitudinal arch, basic gait parameters and balance."

ELIGIBILITY:
Inclusion Criteria:

- Bilateral flexible flatfeet

Exclusion Criteria:

* Tarsal coalitions,
* Congenital defects of the lower limbs,
* Neurological diseases,
* Previous foot surgery.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Navicular Height (NH) | Baseline
  The localization of the medial navicular tuberosity and its distance from the floor as NH will be done in a standing position. The result will be given in millimeters.
Navicular Height (NH) | 6-weeks intervention
  The localization of the medial navicular tuberosity and its distance from the floor as NH will be done in a standing position. The result will be given in millimeters.
Navicular Height (NH) | 3 months later
  The localization of the medial navicular tuberosity and its distance from the floor as NH will be done in a standing position. The result will be given in millimeters.
Navicular Height (NH) | 6 months later
  The localization of the medial navicular tuberosity and its distance from the floor as NH will be done in a standing position. The result will be given in millimeters.
Body Mass Index (BMI) | baseline
  Each child's weight and height will be assessed to determine their BMI using the formula weight [kg] / height [m] 2.
  This will be interpreted according to the international cut-off points. In addition, body composition will be analyzed using bioelectric impedance.
Body Mass Index (BMI) | 6-weeks intervention
  Each child's weight and height will be assessed to determine their BMI using the formula weight [kg] / height [m] 2.
  This will be interpreted according to the international cut-off points. In addition, body composition will be analyzed using bioelectric impedance.
Body Mass Index (BMI) | 3 months later
  Each child's weight and height will be assessed to determine their BMI using the formula weight [kg] / height [m] 2.
  This will be interpreted according to the international cut-off points. In addition, body composition will be analyzed using bioelectric impedance.
Body Mass Index (BMI) | 6 months later
  Each child's weight and height will be assessed to determine their BMI using the formula weight [kg] / height [m] 2.
  This will be interpreted according to the international cut-off points. In addition, body composition will be analyzed using bioelectric impedance.

SECONDARY OUTCOMES:
Foot Posture Index-6 (FPI-6) | Baseline
  The FPI-6 scale consists of 6 separate grades that are then summarized to give a score that reflects foot position. The scale makes it possible to analyze the entire FPI-6 result, as well as to consider the results for individual components. Each of the six parts of FPI-6 is rated on a scale of -2 to +2. The neutral position of the foot is classified as 0, during which pronation becomes positive and supination negative.
Foot Posture Index-6 (FPI-6) | 6-weeks intervention
  The FPI-6 scale consists of 6 separate grades that are then summarized to give a score that reflects foot position. The scale makes it possible to analyze the entire FPI-6 result, as well as to consider the results for individual components. Each of the six parts of FPI-6 is rated on a scale of -2 to +2. The neutral position of the foot is classified as 0, during which pronation becom
Foot Posture Index-6 (FPI-6) | 3 months later
  The FPI-6 scale consists of 6 separate grades that are then summarized to give a score that reflects foot position. The scale makes it possible to analyze the entire FPI-6 result, as well as to consider the results for individual components. Each of the six parts of FPI-6 is rated on a scale of -2 to +2. The neutral position of the foot is classified as 0, during which pronation becomes positive and supination negative
Foot Posture Index-6 (FPI-6) | 6 months later
  The FPI-6 scale consists of 6 separate grades that are then summarized to give a score that reflects foot position. The scale makes it possible to analyze the entire FPI-6 result, as well as to consider the results for individual components. Each of the six parts of FPI-6 is rated on a scale of -2 to +2. The neutral position of the foot is classified as 0, during which pronation becomes positive and supination negative.
Arch Index (AI) | baseline
  The AI will be calculated from a footprint, which clearly defines the weightbearing area of the foot. The footprint will be marked with a "foot axis" line from the centre of the heel to the second toe. The foot axis line will be then separated into 3 equal sections with the separated areas defined as A (forefoot), B (midfoot), and C (rearfoot). This process follows that reported by Cavanagh and Rodgers. The Arch Index (AI) will be obtained from the formula B/A+B+C with the weightbearing area of the toes excluded from the calculation of the AI ratio.
Arch Index (AI) | 6-weeks intervention
  The AI will be calculated from a footprint, which clearly defines the weightbearing area of the foot. The footprint will be marked with a "foot axis" line from the centre of the heel to the second toe. The foot axis line will be then separated into 3 equal sections with the separated areas defined as A (forefoot), B (midfoot), and C (rearfoot). This process follows that reported by Cavanagh and Rodgers. The Arch Index (AI) will be obtained from the formula B/A+B+C with the weightbearing area of the toes excluded from the calculation of the AI ratio.
Arch Index (AI) | 3 months later
  The AI will be calculated from a footprint, which clearly defines the weightbearing area of the foot. The footprint will be marked with a "foot axis" line from the centre of the heel to the second toe. The foot axis line will be then separated into 3 equal sections with the separated areas defined as A (forefoot), B (midfoot), and C (rearfoot). This process follows that reported by Cavanagh and Rodgers. The Arch Index (AI) will be obtained from the formula B/A+B+C with the weightbearing area of the toes excluded from the calculation of the AI ratio.
Arch Index (AI) | 6 months later
  The AI will be calculated from a footprint, which clearly defines the weightbearing area of the foot. The footprint will be marked with a "foot axis" line from the centre of the heel to the second toe. The foot axis line will be then separated into 3 equal sections with the separated areas defined as A (forefoot), B (midfoot), and C (rearfoot). This process follows that reported by Cavanagh and Rodgers. The Arch Index (AI) will be obtained from the formula B/A+B+C with the weightbearing area of the toes excluded from the calculation of the AI ratio.
VICON | baseline
  "Vicon Nexus gait analysis system with 10 Cameras MX-T20 and with three AMTI platforms sampled at 1000 Hz will be used to capture foot kinematics during barefoot walking and self-selected speed along 14m walkway. Markers will be placed according to the Oxford Foot Model (OFM) and the Lower body Plug-in gait Model (PIG) sampled at 200 Hz.
  The data will be repeated until 5 clean completed passes. The Data will then be imported into Poligon 3D motion of the hindfoot to tibia, forefoot to hindfoot, as well as hallux to forefoot and the arch height will be extracted according to the OFM . For each foot, kinematic and kinetic traces will be checked visually and inconsistent trials will be removed."
VICON | 6-weeks intervention
  "Vicon Nexus gait analysis system with 10 Cameras MX-T20 and with three AMTI platforms sampled at 1000 Hz will be used to capture foot kinematics during barefoot walking and self-selected speed along 14m walkway. Markers will be placed according to the Oxford Foot Model (OFM) and the Lower body Plug-in gait Model (PIG) sampled at 200 Hz.
  The data will be repeated until 5 clean completed passes. The Data will then be imported into Poligon 3D motion of the hindfoot to tibia, forefoot to hindfoot, as well as hallux to forefoot and the arch height will be extracted according to the OFM . For each foot, kinematic and kinetic traces will be checked visually and inconsistent trials will be removed."
VICON | 3 months later
  "Vicon Nexus gait analysis system with 10 Cameras MX-T20 and with three AMTI platforms sampled at 1000 Hz will be used to capture foot kinematics during barefoot walking and self-selected speed along 14m walkway. Markers will be placed according to the Oxford Foot Model (OFM) and the Lower body Plug-in gait Model (PIG) sampled at 200 Hz.
  The data will be repeated until 5 clean completed passes. The Data will then be imported into Poligon 3D motion of the hindfoot to tibia, forefoot to hindfoot, as well as hallux to forefoot and the arch height will be extracted according to the OFM . For each foot, kinematic and kinetic traces will be checked visually and inconsistent trials will be removed."
VICON | 6 months later
  "Vicon Nexus gait analysis system with 10 Cameras MX-T20 and with three AMTI platforms sampled at 1000 Hz will be used to capture foot kinematics during barefoot walking and self-selected speed along 14m walkway. Markers will be placed according to the Oxford Foot Model (OFM) and the Lower body Plug-in gait Model (PIG) sampled at 200 Hz.
  The data will be repeated until 5 clean completed passes. The Data will then be imported into Poligon 3D motion of the hindfoot to tibia, forefoot to hindfoot, as well as hallux to forefoot and the arch height will be extracted according to the OFM . For each foot, kinematic and kinetic traces will be checked visually and inconsistent trials will be removed."
BIODEX | baseline
  Biodex Balance System SD 115VAC will be used as equipment for testing static and dynamic stability. Dynamic posture assessment will be performed on the unstable platform using the test on level 5 and 12 to 8 (12 as the most stable platform, 1 the least). Familiarization with the test procedure will be performed prior to the test. The patient's data: age, height and the position of feet in relation to the third metatarsal bone as well as the heel position will be entered into the platform. Three indicators will be obtained: AP - anterior/posterior, ML - medial/lateral and OSI - overall stability index. During the evaluation each child will be asked to stand in the centre of the platform bare feet with arms along the body, looking straight ahead, focusing on the visual feedback screen. For each level of the dynamic stability measurement three trials will be performed and the average will be calculated. Children will be tested in two conditions: with eyes open and closed.
BIODEX | 6-weeks intervention
  Biodex Balance System SD 115VAC will be used as equipment for testing static and dynamic stability. Dynamic posture assessment will be performed on the unstable platform using the test on level 5 and 12 to 8 (12 as the most stable platform, 1 the least). Familiarization with the test procedure will be performed prior to the test. The patient's data: age, height and the position of feet in relation to the third metatarsal bone as well as the heel position will be entered into the platform. Three indicators will be obtained: AP - anterior/posterior, ML - medial/lateral and OSI - overall stability index. During the evaluation each child will be asked to stand in the centre of the platform bare feet with arms along the body, looking straight ahead, focusing on the visual feedback screen. For each level of the dynamic stability measurement three trials will be performed and the average will be calculated. Children will be tested in two conditions: with eyes open and closed.
BIODEX | 3 months later
  Biodex Balance System SD 115VAC will be used as equipment for testing static and dynamic stability. Dynamic posture assessment will be performed on the unstable platform using the test on level 5 and 12 to 8 (12 as the most stable platform, 1 the least). Familiarization with the test procedure will be performed prior to the test. The patient's data: age, height and the position of feet in relation to the third metatarsal bone as well as the heel position will be entered into the platform. Three indicators will be obtained: AP - anterior/posterior, ML - medial/lateral and OSI - overall stability index. During the evaluation each child will be asked to stand in the centre of the platform bare feet with arms along the body, looking straight ahead, focusing on the visual feedback screen. For each level of the dynamic stability measurement three trials will be performed and the average will be calculated. Children will be tested in two conditions: with eyes open and closed.
BIODEX | 6 months later
  Biodex Balance System SD 115VAC will be used as equipment for testing static and dynamic stability. Dynamic posture assessment will be performed on the unstable platform using the test on level 5 and 12 to 8 (12 as the most stable platform, 1 the least). Familiarization with the test procedure will be performed prior to the test. The patient's data: age, height and the position of feet in relation to the third metatarsal bone as well as the heel position will be entered into the platform. Three indicators will be obtained: AP - anterior/posterior, ML - medial/lateral and OSI - overall stability index. During the evaluation each child will be asked to stand in the centre of the platform bare feet with arms along the body, looking straight ahead, focusing on the visual feedback screen. For each level of the dynamic stability measurement three trials will be performed and the average will be calculated. Children will be tested in two conditions: with eyes open and closed.
Y-BALANCE TEST | baseline
  The children will be acquainted with the methodology of the test and testing procedures. Prior to formal testing children will practise 6 trials on each leg in 3 reach directions. The children will perform one leg stand in the centre of the grid, with the most distal aspect of the great toe at the starting line. While maintaining a single-leg stance, the children will be asked to reach the anterior, posteromedial and posterolateral directions with the lifted limb. The whole process will be repeated while standing on the other leg. The maximal reaching point will be considered for the future analysis. The trial will be discarded and repeated if the children (1) fail to maintain unilateral stance, (2) lift or move the stance foot from the grid, (3) touch down with the reach foot, or (4) fail to return the reach foot to the starting position. Three proper trials in each reach direction will be used for analysis.
Y-BALANCE TEST | 6-weeks intervention
  The children will be acquainted with the methodology of the test and testing procedures. Prior to formal testing children will practise 6 trials on each leg in 3 reach directions. The children will perform one leg stand in the centre of the grid, with the most distal aspect of the great toe at the starting line. While maintaining a single-leg stance, the children will be asked to reach the anterior, posteromedial and posterolateral directions with the lifted limb. The whole process will be repeated while standing on the other leg. The maximal reaching point will be considered for the future analysis. The trial will be discarded and repeated if the children (1) fail to maintain unilateral stance, (2) lift or move the stance foot from the grid, (3) touch down with the reach foot, or (4) fail to return the reach foot to the starting position. Three proper trials in each reach direction will be used for analysis.
Y-BALANCE TEST | 3 months later
  The children will be acquainted with the methodology of the test and testing procedures. Prior to formal testing children will practise 6 trials on each leg in 3 reach directions. The children will perform one leg stand in the centre of the grid, with the most distal aspect of the great toe at the starting line. While maintaining a single-leg stance, the children will be asked to reach the anterior, posteromedial and posterolateral directions with the lifted limb. The whole process will be repeated while standing on the other leg. The maximal reaching point will be considered for the future analysis. The trial will be discarded and repeated if the children (1) fail to maintain unilateral stance, (2) lift or move the stance foot from the grid, (3) touch down with the reach foot, or (4) fail to return the reach foot to the starting position. Three proper trials in each reach direction will be used for analysis.
Y-BALANCE TEST | 6 months later
  The children will be acquainted with the methodology of the test and testing procedures. Prior to formal testing children will practise 6 trials on each leg in 3 reach directions. The children will perform one leg stand in the centre of the grid, with the most distal aspect of the great toe at the starting line. While maintaining a single-leg stance, the children will be asked to reach the anterior, posteromedial and posterolateral directions with the lifted limb. The whole process will be repeated while standing on the other leg. The maximal reaching point will be considered for the future analysis. The trial will be discarded and repeated if the children (1) fail to maintain unilateral stance, (2) lift or move the stance foot from the grid, (3) touch down with the reach foot, or (4) fail to return the reach foot to the starting position. Three proper trials in each reach direction will be used for analysis.
sEMG | baseline
  "A sixteen-channel sEMG system will be used to recorded muscle activation. The sEMG and acceleration data will be transmitted to computer where the analogue data will be sampled at 2000Hz and stored for analysis.
  The tibialis anterior, peroneus longus, medial and lateral gastrocnemius, abductor hallucis longus sEMG will be recorded with the use of surface electrodes. The application of the surface electrodes will be performed following the SENIAM's recommendations, additional abductor hallucis longus muscle, the sEMG electrodes will be placed approximately 1-2 cm posterior to the navicular tuberosity. The skin at the electrode sites will be properly prepared.
  The sEMG data will be collected in coordination with Vicon data."
sEMG | 6-weeks intervention
  "A sixteen-channel sEMG system will be used to recorded muscle activation. The sEMG and acceleration data will be transmitted to computer where the analogue data will be sampled at 2000Hz and stored for analysis.
  The tibialis anterior, peroneus longus, medial and lateral gastrocnemius, abductor hallucis longus sEMG will be recorded with the use of surface electrodes. The application of the surface electrodes will be performed following the SENIAM's recommendations, additional abductor hallucis longus muscle, the sEMG electrodes will be placed approximately 1-2 cm posterior to the navicular tuberosity. The skin at the electrode sites will be properly prepared.
  The sEMG data will be collected in coordination with Vicon data."
sEMG | 3 months later
  "A sixteen-channel sEMG system will be used to recorded muscle activation. The sEMG and acceleration data will be transmitted to computer where the analogue data will be sampled at 2000Hz and stored for analysis.
  The tibialis anterior, peroneus longus, medial and lateral gastrocnemius, abductor hallucis longus sEMG will be recorded with the use of surface electrodes. The application of the surface electrodes will be performed following the SENIAM's recommendations, additional abductor hallucis longus muscle, the sEMG electrodes will be placed approximately 1-2 cm posterior to the navicular tuberosity. The skin at the electrode sites will be properly prepared.
  The sEMG data will be collected in coordination with Vicon data."
sEMG | 6 months later
  "A sixteen-channel sEMG system will be used to recorded muscle activation. The sEMG and acceleration data will be transmitted to computer where the analogue data will be sampled at 2000Hz and stored for analysis.
  The tibialis anterior, peroneus longus, medial and lateral gastrocnemius, abductor hallucis longus sEMG will be recorded with the use of surface electrodes. The application of the surface electrodes will be performed following the SENIAM's recommendations, additional abductor hallucis longus muscle, the sEMG electrodes will be placed approximately 1-2 cm posterior to the navicular tuberosity. The skin at the electrode sites will be properly prepared.
  The sEMG data will be collected in coordination with Vicon data."

CONTACTS AND LOCATIONS:
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Poland